CLINICAL TRIAL: NCT03664323
Title: Efficacy of Chemotherapy or Chemo-anti-PD-1 Combination After Failed Anti-PD-1 Therapy for Relapsed and Refractory Hodgkin Lymphoma: a Series From Lysa Centers.
Brief Title: Anti-PD-1 and Chemotherapy for R/R Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Anti-PD-1 Hodgkin
Record Dates: First submitted 2018-06-04; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Immunotherapy; chemotherapy; anti-PD1; re-sensibilization
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 Sequential strategy: Patients for whom anti-PD-1 therapy was stopped with the introduction of a new treatment line (19 patients, 63%).
  Interventions: Biological: Evaluate the improvement in response from the end of anti-PD-1 monotherapy
- Group 2 Concomitant strategy: Patients for whom a combination of CT with anti-PD-1 therapy was initiated (11 patients, 37 %).
  Interventions: Biological: Evaluate the improvement in response from the end of anti-PD-1 monotherapy

INTERVENTIONS:
Biological: Evaluate the improvement in response from the end of anti-PD-1 monotherapy — Evaluate the improvement in response from the end of anti-PD-1 monotherapy to the first evaluation after introduction of CT alone (Group 1) or combined with anti-PD-1 (Group 2).

SUMMARY:
Anti-PD-1 therapy provides high response rates in Hodgkin lymphoma (HL) patients who have relapsed or are refractory (R/R) to autologous stem cell transplantation (ASCT) and brentuximab vedotin (BV), but median progression free survival (PFS) is only one year. The efficacy of treatment following anti-PD-1 is not well known.

In this context, the optimal treatment for patients who failed after anti-PD-1 therapy is an issue. To better assess their outcome, the investigators retrospectively analyzed the characteristics and outcome of patients from 14 LYSA (The Lymphoma Study Association) centers who lost response to anti-PD-1 therapy and received additional CT.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of classical HL
* Optional histopathology confirmation of relapse/refractory HL, (2) age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 to 2
* Patients must be have received: at least 2 prior regimens and have received or be ineligible for autologous stem cell transplant and must have received prior BV, and at least 2 cycles of single agent anti-PD-1 as last treatment before entering the study,
* Patients must have inadequate response to anti-PD-1 monotherapy (progressive disease or partial response according to Lugano criteria) with at least one hypermetabolic lesion over the liver and mediastinum background at time of inclusion in the study
* Previous allogeneic stem cell transplant was allowed. Patients treated with radiotherapy alone after anti-PD1 or combined with anti-PD1 treatment were not included in the study.

Exclusion Criteria:

- radiotherapy in the treatment after anti-PD1

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The initial diagnosis of classical HL was established from biopsies in accordance with the 2008 World Health Organization classification14. We retrospectively analyzed 30 R/R classical HL patients from 14 LYSA centers who received anti-PD-1 therapy as part of a clinical trial (n=4), from an off-label program authorization for temporary use (ATU) from the French medical drug agency (Agence Nationale de Sécurité du Médicament, ANSM) (n=22), from the Belgian national system for the reimbursement of health care (Institut National d'Assurance Maladie Invalidité, INAMI) (n=4).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate after re-exposure to chemotherapy | 10 weeks
  Patient evaluation was timed by treating physicians according to the policy of each center, and all patients were evaluated after a median of 10 weeks (min 7 weeks, max 12 weeks) with PET/CT using Lugano criteria

SECONDARY OUTCOMES:
Best response obtained (Group 1) | 10 weeks
  the best response obtained with CT after anti-PD-1
Best response obtained (Group 2) | 10 weeks
  the best response obtained with CT after the combination anti-PD-1 and CT
The toxicities experienced during CT or anti-PD-1 plus CT combination | 10 weeks
  The toxicities were graded retrospectively according to the National Cancer Institute Common Toxicity Criteria for AEs (version 4.0).
Outcomes including PFS | up to 12 months
  PFS was defined as the time from first relapse, or progression, to the next event (defined as either second relapse/progression, change of therapy, or death from any cause)
Outcomes including overall survival (OS). | up to 24 months
  OS was defined as the time from first relapse, or progression, to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé GHESQUIERES, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France